CLINICAL TRIAL: NCT04130997
Title: An Open Label Extension Study of Ublituximab in Subjects With Relapsing Multiple Sclerosis
Brief Title: An Extension Study of Ublituximab in Participants With Relapsing Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG1101-RMS303; 2019-003625-16 (EudraCT Number)
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
MeSH Terms: interventions — ublituximab

STUDY DESIGN:
Intervention Model Description: open-label, single-arm, extension study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ublituximab Infusions (Experimental): RMS301/RMS302: All participants transferring from RMS301/RMS302 who sign consent for this study will receive an initial 4-hour infusion of 150 mg ublituximab on Week 1 (Day 1) followed by a 1-hour infusion of 450 mg ublituximab 14 days later Week 3 (Day 15). Subsequent infusions of ublituximab will be administered at 450 mg for 1-hour every 24 weeks from Weeks 24 to 312.
  RMS201E: All participants transferring from RMS201E who sign consent for this study will receive a 1-hour infusion of 450 mg ublituximab on Week 1 (Day 1) and subsequent infusions of ublituximab will be administered at 450 mg for 1-hour every 24 weeks from Weeks 24 to 312.
  For all participants (RMS301/RMS302/RMS201E), infusion treatment will continue for 312 weeks, or until physician or participant decision to withdraw from the study.
  Interventions: Biological: Ublituximab

INTERVENTIONS:
Biological: Ublituximab — Ublituximab (TG-1101) is a recombinant chimeric monoclonal antibody targeting CD20, available as a 25 mg/mL concentrate for intravenous use, supplied by TG Therapeutics, Inc.
  Other Names: TG-1101

SUMMARY:
The purpose of this study is to evaluate long-term safety and efficacy of ublituximab therapy in participants with relapsing multiple sclerosis (RMS).

DETAILED DESCRIPTION:
TG1101-RMS303 is an open-label, single-arm extension study designed to evaluate long-term safety and efficacy of ublituximab in participants with RMS. Participants who complete the 96-week, double-blind treatment period of TG1101-RMS301 (RMS301 [NCT03277261]) or TG1101-RMS302 (RMS302 [NCT03277248]) are eligible for participation in this Open Label Extension (OLE) study. Participants may also be eligible for TG1101-RMS303 if they have completed Week 208 of TG1101-RMS201E (RMS201E [NCT03381170]) (United States of America [USA] participants only).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria:

1. Complete the 96-week double-blind TG1101-RMS301 (NCT03277261) or TG1101-RMS302 (NCT03277248) study or complete the final Week 208 visit of the TG1101-RMS201E (NCT03381170) study
2. Investigator believes may benefit from treatment with ublituximab
3. Are able and willing to provide written informed consent (e.g., before the first infusion) and to comply with the study protocol
4. Female participants of child-bearing potential, and male partners must consent to use a medically acceptable method of contraception from consent, throughout the study period, and for 20 weeks after the last dose of ublituximab

Exclusion Criteria:

Participants who meet any of the following exclusion criteria are not to be enrolled to this study:

1. Any significant or uncontrolled medical condition or treatment-emergent, clinically significant laboratory abnormality such as:

   1. Absolute neutrophil count < 1.5 x 10e3/µL
   2. Hematocrit < 24%
   3. Platelet count < 150,000 cell/mm^3
   4. Hypogammaglobulinemia immunoglobulin G (IgG) < 4.0g/L
2. Active infection
3. Ongoing pregnancy (female participants)
4. Participants who discontinued ublituximab treatment or withdrew consent from the TG1101-RMS301 or TG1101-RMS302 study during the 96-week evaluation period or prior to completing the final Week 208 visit of the TG1101-RMS201E study
5. Participants who have started any disease modifying therapy (DMT), stem cell transplantation, or participation in any other interventional clinical trial after completion of the 96-week visit in the TG1101-RMS301, TG1101-RMS302, or after completing the final Week 208 visit of the TG1101-RMS201E study
6. Participants who have had a confirmed multiple sclerosis (MS) relapse within the past 30 days prior to Week 1 Day 1 (W1D1). Following a relapse, participants must be neurologically stable for at least 30 days prior to screening or W1D1 of the OLE
7. Participants with unstable disease activity
8. Presence of malignancy, except for surgically excised basal or squamous cell skin lesions
9. Vaccination with live virus within 2 months of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | Up to Week 336
  ARR is defined as the number of relapses per-participant year. The estimate of ARR will be the total number of relapses divided by the sum of duration on study treatment (years).

CONTACTS AND LOCATIONS:
Locations (66):
- United States (19):
  - TG Therapeutics Investigational Trial Site, Pasadena, California
  - TG Therapeutics Investigational Trial Site, Denver, Colorado
  - TG Therapeutics Investigational Trial Site, Miami, Florida
  - TG Therapeutics Investigational Trial Site, Tampa, Florida
  - TG Therapeutics Investigational Trial Site, Northbrook, Illinois
  - TG Therapeutics Investigational Trial Site, Kansas City, Kansas
  - TG Therapeutics Investigational Trial Site, Detroit, Michigan
  - TG Therapeutics Investigational Trial Site, Las Vegas, Nevada
  - TG Therapeutics Investigational Trial Site, Teaneck, New Jersey
  - TG Therapeutics Investigational Trial Site, Albuquerque, New Mexico
  - TG Therapeutics Investigational Trial Site, Amherst, New York
  - TG Therapeutics Investigational Trial Site, Columbus, Ohio
  - TG Therapeutics Investigational Trial Site, Westerville, Ohio
  - TG Therapeutics Investigational Trial Site, Knoxville, Tennessee
  - TG Therapeutics Investigational Trial Site, Dallas, Texas
  - TG Therapeutics Investigational Trial Site, Frisco, Texas
  - TG Therapeutics Investigational Trial Site, Round Rock, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas
  - TG Therapeutics Investigational Trial Site, Seattle, Washington
- Belarus (2):
  - TG Therapeutics Investigational Trial Site, Grodno
  - TG Therapeutics Investigational Trial Site, Minsk
- Croatia (3):
  - TG Therapeutics Investigational Trial Site, Osijek
  - TG Therapeutics Investigational Trial Site, Varaždin
  - TG Investigational Trial Site, Zagreb
- TG Therapeutics Investigational Trial Site, Tbilisi, Georgia
- Poland (7):
  - TG Therapeutics Investigational Trial Site, Katowice
  - TG Therapeutics Investigational Trial Site, Krakow
  - TG Therapeutics Investigational Trial Site, Lodz
  - TG Therapeutics Investigational Trial Site, Olsztyn
  - TG Therapeutics Investigational Trial Site, Poznan
  - TG Therapeutics Investigational Trial Site, Warsaw
  - TG Therapeutics Investigational Trial Site, Zabrze
- Russia (18):
  - TG Therapeutics Investigational Trial Site, Arkhangelsk
  - TG Therapeutics Investigational Trial Site, Barnaul
  - TG Therapeutics Investigational Trial Site, Bryansk
  - TG Therapeutics Investigational Trial Site, Chelyabinsk
  - TG Therapeutics Investigational Trial Site, Kemerovo
  - TG Therapeutics Investigational Trial Site, Krasnoyarsk
  - TG Therapeutics Investigational Trial Site, Kursk
  - TG Therapeutics Investigational Trial Site, Moscow
  - TG Therapeutics Investigational Trial Site, Nizhny Novgorod
  - TG Therapeutics Investigational Trial Site, Novosibirsk
  - TG Therapeutics Investigational Trial Site, Pyatigorsk
  - TG Therapeutics Investigational Trial Site, Saint Petersburg
  - TG Therapeutics Investigational Trial Site, Saransk
  - TG Therapeutics Investigational Trial Site, Smolensk
  - TG Therapeutics Investigational Trial Site, Tomsk
  - TG Therapeutics Investigational Trial Site, Tyumen
  - TG Therapeutics Investigational Trial Site, Ufa
  - TG Therapeutics Investigational Trial Site, Yekaterinburg
- Serbia (2):
  - TG Therapeutics Investigational Trial Site, Belgrade
  - TG Therapeutics Investigational Trial Site, Kragujevac
- Ukraine (14):
  - TG Therapeutics Investigational Trial Site, Cherkasy
  - TG Therapeutics Investigational Trial Site, Chernihiv
  - TG Therapeutics Investigational Trial Site, Chernivtsi
  - TG Therapeutics Investigational Trial Site, Ivano-Frankivsk
  - TG Therapeutics Investigational Trial Site, Kharkiv
  - TG Therapeutics Investigational Trial Site, Kyiv
  - TG Therapeutics Investigational Trial Site, Lviv
  - TG Therapeutics Investigational Trial Site, Odesa
  - TG Therapeutics Investigational Trial Site, Poltava
  - TG Therapeutics Investigational Trial Site, Ternopil
  - TG Therapeutics Investigational Trial Site, Uzhhorod
  - TG Therapeutics Investigational Trial Site, Vinnytsia
  - TG Therapeutics Investigational Trial Site, Zaporizhia
  - TG Therapeutics Investigational Trial Site, Zhytomyr